CLINICAL TRIAL: NCT05494554
Title: Comparison of Mechanical Power Calculations of Volume Control and Pressure Control Modes: A Prospective Observational Study
Brief Title: Comparison of Mechanical Power Calculations of Volume Control and Pressure Control Modes
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-02-23
Record Dates: First submitted 2022-07-21; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pressure control mode group: On the 2nd day of intensive care hospitalization, while under deep sedation and in the controlled mode (VCV or PRVC) and in the supine position, the ventilator in the VCV mode was switched to PRVC mode for 60 minutes without changing any of the set ventilator settings (RR, PEEP, TV, I:E ratio).
  Interventions: Device: Changing mechanical ventilation mode
- Volume control mode group: Likewise, if it is in PRVC mode, it is also switched to VCV mode for 60 minutes. In this way, two dependent groups were formed.
  Interventions: Device: Changing mechanical ventilation mode

INTERVENTIONS:
Device: Changing mechanical ventilation mode — On the 2nd day of intensive care hospitalization, while under deep sedation and in the controlled mode (VCV or PRVC) and in the supine position, the ventilator in the VCV mode was switched to PRVC mode for 60 minutes without changing any of the set ventilator settings (RR, PEEP, TV, I:E ratio). Likewise, if it is in PRVC mode, it is also switched to VCV mode for 60 minutes. MP values were calculated from the minute respiratory parameters of all patients with the MP formulas defined in the software.

SUMMARY:
The management of ARDS, which is one of the important problems of intensive care patients, has gained popularity with the pandemic. Mechanical ventilation is an important life-saving treatment in ARDS patients. However, when not used correctly, it can cause Ventilator-Induced Lung Injury (VILI). Therefore, lung protective ventilation should be applied to minimize VILI in ARDS patients. Mechanical power is one of the parameters that guides intensivist in predicting VILI.

DETAILED DESCRIPTION:
The goal of mechanical ventilation in ARDS patients is to improve oxygenation by reducing the work of breathing . With this aim, the orientation towards sensitive ventilation strategies has increased in the light of experience and scientific data from the past to the present. Today, the concept of Mechanical Power (MP) has been developed, which combines different variables, such as tidal volume, drive pressure, gas flow, respiratory rate, and PEEP, which have been associated with VILI in various studies, into a single parameter. In this study, the investigators used the simplified MP equation (MPvcv (simpl)) developed by Gattinoni et al. for power calculation in volume control mode and the simplified MP equation (MPpcv(simpl)) developed by Becher et al. for power calculation in pressure control mode. Thus, the investigators aimed to compare the volume control and pressure control modes over the concept of MP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Covid-19 diagnosis in intensive care unit (ICU) and diagnosed with ARDS according to Berlin criteria
* Intubated patients which treated in the supine position on the second day of ICU admission

Exclusion Criteria:

* Patients with a known diagnosis of COPD
* Patients experiencing hemodynamic instability during ventilation
* Prone pozisyonda olan hastalar
* Patients receiving inotropic support
* Patients with missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted prospectively with 36 Covid-19 ARDS patients who were followed up in the Dr. Sadi Konuk Training and Research Hospital Anesthesia and Intensive Care Unit and diagnosed with ARDS according to the Berlin criteria. The definite COVID-19 diagnosis was confirmed by PCR (Bio-Speedy Covid-19 RT-Qpcr detection Kit-Bioeksen, Turkey) obtained from the nasal swab sample and chest computed tomography images.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-01-22 (Actual)

PRIMARY OUTCOMES:
Mechanical power values of different ventilation modes | 60 minutes
  We aimed to compare the volume control and pressure control modes over the mechanical power values.

CONTACTS AND LOCATIONS:
Overall Officials: Furkan Tontu, Principal Investigator — Intensivist
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided